CLINICAL TRIAL: NCT06013748
Title: Virtual Reality Therapy for Voice Hearing (VR-VOICES): a Randomized Controlled Trial
Acronym: VR-VOICES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL78885.042.22; 60-63600-98-1055 / 636320017 (Other Grant/Funding Number: ZonMW)
Record Dates: First submitted 2023-07-18; First posted 2023-08-28 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Hallucinations, Verbal Auditory
Keywords: Virtual reality; Auditory hallucination; Voice-hearing; Psychological intervention
MeSH Terms: conditions — Hallucinations | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VR-VOICES (Experimental): 7-10 sessions of 45-60 minutes of individual VR assisted therapy and two booster sessions, in addition to TAU. Participants allocated to VR-VOICES create together with their therapist a VR digital representation (avatar with face, body and voice) of the voice that bothers them most. Patients have dialogues with the avatar, voiced by the therapist. As indicated in the treatment protocol, over the sessions the avatar will become less hostile and the participant will gain more power and resilience over the avatar.
  Interventions: Behavioral: VR-VOICES
- Treatment as usual (Other): TAU as described in the current Dutch treatment guidelines, which generally exists of pharmacological treatment, supportive counseling, and psychological interventions such as CBT and coping strategies. This will vary per individual.
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: VR-VOICES — 7-10 individual VR assisted therapy for voice-hearing session and two booster sessions, in addition to TAU.
  Arms: VR-VOICES
Other: Treatment as usual — Treatment as usual as provided by the mental health centers
  Arms: Treatment as usual

SUMMARY:
Rationale: Auditory verbal hallucinations (AVH) - hearing voices that others cannot hear - are common in mental illnesses. For many people AVH are distressing, disabling and persistent, despite medication. Current psychological interventions show low to medium effects. Preliminary studies suggest that an innovative empowering psychological therapy using computer simulations representing the AVH (avatars) can be effective for reducing AVH distress and frequency. Virtual reality (VR) has the potential to improve this treatment. Therefore, we developed a novel VR treatment for this problem. In this study, the effect of this treatment will be investigated.

Objective: To test the effect of a novel VR treatment for AVH (VR-VOICES) on distress and frequency of AVH in patients with a psychiatric disorder. Furthermore, to investigate the effect of VR-VOICES on clinical symptoms, quality of life, and healthcare costs of the treatment.

DETAILED DESCRIPTION:
Study design: Single-blind randomized controlled intervention trial (RCT) with two arms: VR-VOICES as intervention and treatment as usual (TAU) as a control condition.

Study population: Patients with a DSM-5 diagnosis who have experienced distressing AVH for at least 3 months, who are 16 years or older (N=112).

Intervention:

* VR-VOICES intervention: 7-10 sessions of 45-60 minutes of individual VR assisted therapy and two booster sessions, in addition to TAU. Participants allocated to VR-VOICES create together with their therapist a VR digital representation (avatar with face, body and voice) of the voice that bothers them most. Patients have dialogues with the avatar, voiced by the therapist. As indicated in the treatment protocol, over the sessions the avatar will become less hostile and the participant will gain more power and resilience over the avatar.
* Control: TAU as described in the current Dutch treatment guidelines, which generally exists of pharmacological treatment, supportive counseling, and psychological interventions such as CBT and coping strategies.

Main study parameters/endpoints: Assessments will be obtained at baseline, within some VR-VOICES sessions, posttreatment (12 weeks after baseline), and at 6-month follow-up. Primary outcome: severity of AVH (total score on the auditory hallucinations scale of the PSYRATS) at post-treatment. Secondary outcomes: in-depth characteristics of AVH such as the frequency, voice impact, beliefs about voices, power relative to voices, levels of anxiety, distress and impact on daily life as measured with questionnaires and diary assessments in the flow of daily life. Other secondary outcomes include clinical symptoms, cost-effectiveness and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Having a DSM-5 diagnosis of a psychiatric disorder
* Distressing AVH for minimally 3 months.
* Age 16 years or older

Exclusion Criteria:

* Insufficient command of the Dutch language
* Unable to provide informed consent
* Primary diagnosis of a substance use disorder, or organic brain disease (such as dementia)
* A degree of substance abuse that hinders treatment adherence
* Auditory verbal hallucinations in a language not spoken by therapists
* Patients cannot receive CBT specifically focused at gaining empowerment over voices during the study period or 6 months prior to enrolment.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2022-10-31 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Voices severity | Between baseline and posttreatment after 3 months
  The Psychotic Symptoms Rating Scales (PSYRATS) is a semi-structured interview to assess characteristics of hallucinations and delusions. The auditory hallucinations subscale (AHS), which is used as the primary outcome, has 11 items.

SECONDARY OUTCOMES:
Voice severity (frequency and distress) and delusions | Assessment at baseline, 3 months (posttreatment), 6 months (follow-up)
  The Psychotic Symptoms Rating Scales (PSYRATS) is a semi-structured interview to assess characteristics of hallucinations and delusions. The auditory hallucinations subscale (AHS) has 11 items.The delusions subscale (DS) has six items.
Beliefs about voice power, voice intent and responding styles (Beliefs about Voices Questionnaire-Revised, BAVQ-R) | Assessment at baseline, 3 months (posttreatment), 6 months (follow-up)
  The BAVQ-R has 54 items, measured on a four-point scale: "disagree" (0), "unsure" (1), "slightly agree" (2), "strongly agree"(3).
Social comparison with voices (Social Comparison Rating Scale To Voices, SCRS) | Assessment at baseline, 3 months (posttreatment), 6 months (follow-up)
  The SCRS has 11 items measuring characteristics of the participants as compared to their voices on a 10-point likert scale ranging from 1-10.
Impact of voice-hearing (Voice Impact Scale, VIS) | Assessment at baseline, 3 months (posttreatment), 6 months (follow-up)
  The VIS has 24 items measured on a 10-point likert scale ranging from 1 (totally disagree) to 10 (totally agree).
Voices acceptance (Voices Acceptance and Action scale, VAAS) | Assessment at baseline, 3 months (posttreatment), 6 months (follow-up)
  Section A of the VAAS has 12 items and section B 27. Items are rated on a 5-point scale: strongly disagree, disagree, unsure or neutral, or strongly agree.
Depressive symptoms (Inventory of Depressive Symptomatology, IDS) | Assessment at baseline, 3 months (posttreatment), 6 months (follow-up)
  The IDS-SR is a 30-item questionnaire. Each item has four statements that reflect various degrees of symptom severity, scored on a four-point scale from 0 to 3.
Paranoid ideation (Revised Green Paranoid Thoughts Scale, R-GPTS) | Assessment at baseline, 3 months (posttreatment), 6 months (follow-up)
  The R-GPTS part A consists of 8 items, and B of 10 items. Items are rated on a 5-point scale ranging from 0 (not at all) to 4 (totally).
Self-esteem (Self Esteem Rating Scale, SERS) | Assessment at baseline, 3 months (posttreatment), 6 months (follow-up)
  The SERS has 20 items which are rated on a 7-point likert scale from 1 (strongly disagree) -7 (strongly agree).
Health care costs (Treatment Inventory of Costs in Patients with psychiatric disorders, TIC-P) | Assessment at baseline, 3 months (posttreatment), 6 months (follow-up)
  The TiC-P is a self-report questionnaire that consists of two parts. The first part includes 38 structured questions, starting with yes/no questions and followed by a question on the volume of medical consumption.
Costs production losses (Treatment Inventory of Costs in Patients with psychiatric disorders, TIC-P) | Assessment at baseline, 3 months (posttreatment), 6 months (follow-up)
  The TiC-P is a self-report questionnaire that consists of two parts. The second part deals with 12 questions about work to collect data on productivity losses due to health problems.
Quality of life (Sheehan Disability Scale, SDS) | Assessment at baseline, 3 months (posttreatment), 6 months (follow-up)
  The SDS is a brief, 5-item self-report tool that assesses functional impairment in work/school, social life, and family life on a scale from 0-10, and assess how many days someone missed work/school/responsibilities and how many days someone was unproductive.
Quality of life (EuroQol, EQ-5D-5L) | Assessment at baseline, 3 months (posttreatment), 6 months (follow-up)
  The first 25 items of this questionnaires are based on five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The patient is asked to indicate their health status by choosing the most appropriate level: no problems, slight problems, moderate problems, severe problems, and extreme problems. The last question indicates their current health status on a scale from 0 to 100.
Empowerment/self-efficacy (Mental Health Confidence Scale, MHCS) | Assessment at baseline, 3 months (posttreatment), 6 months (follow-up)
  The MHCS has 16 items that are measured on a 6-point likert scale ranging from totally not confidant
Experience sampling method (ESM) of auditory hallucinations and mental states | Assessment at baseline, 3 months (posttreatment), 6 months (follow-up)
  ESM of auditory verbal hallucinations and mental states measured in the flow of daily life. ESM is a structured diary method for reporting momentary experiences 18. Individuals complete short questionnaires on their mobile device, by pressing a link in a text message. Participants will complete ESM 5x daily for 7 days, completion takes ±1 minute. Participants have to complete the questionnaire within 30 minutes after the text message notification, the interval between measurements is 3 hours.

OTHER OUTCOMES:
Trauma (Trauma and Life Events TALE) | Assessment at baseline
  21 items on traumatic events, whether they happened, more than once and at which age.
Trauma impact (Trauma screening questionnaire (TSQ) | Assessment at baseline
  10 items to screen trauma which can be answered with yes or no.
Medication use | Assessment at baseline, 3 months (posttreatment), 6 months (follow-up)
  Use of prescribed medication in the past 3 months, type of medication, were the medication is for, how often it was used and what amount (in milligram)
Substance use | Assessment at baseline, 3 months (posttreatment), 6 months (follow-up)
  Use of substances, number of glasses of alcohol in the past month. Use of softdrugs and harddrugs in the past 3 months, type of drugs, how often the drugs were used, how much was used each time.
Frequency and type of interventions and training (questionnaire interventions and training) | Assessment at baseline, 3 months (posttreatment), 6 months (follow-up)
  Frequency of use of 21 types of psychological interventions and training in the past 30 days. There is also an option 'other', where specific other interventions and the frequency can be noted down.
Working alliance VR-VOICES (Working Alliance Inventory,WAV) | Assessment at the end of VR-VOICES session 7 (only for the VR-VOICES group), which will be between 7and 10 weeks after baseline is completed.
  The WAV has 36 items for the participant and 36 items for the therapist. Items are rated on a 5-point scale ranging from ''never'' to ''always''
Presence in VR ((Igroup Presence Questionnaire, IPQ) | Assessment during VR-VOICES session 3 & 7 (only for the VR-VOICES group), , which will be between 3-7 weeks (for session 3) and 7-10 weeks (for session 7) after baseline is completed.
  The IPQ has 14 items rated on 7-point likert scale ranging from fully disagree to fully agree.
Fit of avatar and voice. | Assessment during VR-VOICES session 7 (only for the VR-VOICES group), which will be between 7and 10 weeks after baseline is completed.
  Experience of fit of the voice and avatar to the actual voice (two single items on a scale from 1-100).
Session information | Assessment during each VR-VOICES therapy session (only VR-VOICES group), between baseline and 3 months (follow-up)
  Frequency and duration of use of the session recordings by the participant, duration, protocol deviations
Interview VR-VOICES | The interview takes place at 6 months (follow-up) and concerns the experience of the therapy
  After the VR-VOICES intervention, in-depth interviews will be performed to collect the experiences of patients with VR-VOICES. This will be done in a subsample of participants (n=20)

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - Lentis, Groningen, Provincie Groningen
  - GGZ Drenthe, Assen
  - University Medical Center Groningen, Groningen

IPD SHARING:
Plan to Share IPD: No